CLINICAL TRIAL: NCT00130546
Title: A Prospective, Randomized Intra-Individual Study With the Sirolimus Coated Cypher Select(TM) and the Paclitaxel(TM) Coated Express Balloon Expandable Stents for the Treatment of Patients With Two de Novo Native Coronary Artery Lesions.
Brief Title: Intra-Individual Comparison of Sirolimus and Paclitaxel Coated Stent (FRE-RACE Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: Cordis Medizinische Apparate GmbH (Other)
Responsible Party: Prof. Dr. Zehender, University Hospital Freiburg
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FreRace-Study 186/02
Record Dates: First submitted 2005-08-11; First posted 2005-08-15 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; coronary intervention; drug eluting stent implantation; Cypher - Stent; Sirolimus; Taxus - Stent; Paclitaxel
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Cypher Stent
  Interventions: Device: Sirolimus eluting Cypher Select(TM)
- 2 (Active Comparator): Taxus Stent
  Interventions: Device: Paclitaxel-eluting TAXUS(TM)

INTERVENTIONS:
Device: Paclitaxel-eluting TAXUS(TM) — TAXUS(TM) Paclitaxel-eluting stent
  Arms: 2
Device: Sirolimus eluting Cypher Select(TM) — Sirolimus eluting Cypher Select(TM) stent
  Arms: 1

SUMMARY:
The main objective of this study is to assess the safety and effectiveness of the Sirolimus eluting Cypher Select(TM) stent in reducing angiographic in-stent late loss in de novo native coronary lesions as compared to the TAXUS(TM) Paclitaxel-eluting stent in patients presenting with two or more coronary artery stenoses (prospective, randomized, intra-individual comparison).

DETAILED DESCRIPTION:
This is a prospective, 2 arm, randomized, multicenter Phase III study (6 centers).

A total of 110 patients with at least two de novo native coronary artery lesions (lesion A, lesion B) ≤ 30 mm in length and ≥ 2.25 mm to < 3.0 mm in diameter by visual estimate will be enrolled. Patients will be randomized for implantation of the sirolimus eluting Cypher Select(TM) Balloon-Expandable Stent or to the TAXUS(TM) Paclitaxel-eluting stent for lesion A and B.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be >=18 and <=85 years of age
* Female of childbearing potential must have a negative pregnancy test at the time of enrolment and utilize reliable birth control for the duration of their participation in the trial
* Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II-III) and documented ischemia OR patients with documented silent ischemia
* Two or more de novo lesions < 30 mm in length (visual estimate)
* Target vessel at lesion site is ≥ 2.25 mm and ≤ 3.0 mm in diameter (visual estimate)
* Target lesion is located in a native coronary artery which can be covered by one stent (single lesion)
* Acceptable candidate for coronary artery bypass surgery (CABG)
* Target lesion stenosis is > 50% and < 100% (thrombolysis in myocardial infarction [TIMI] 1) (visual estimate)
* Target lesions do not differ in length for more than 6 mm
* Patient is willing to comply with the specified follow-up evaluation
* Patient must provide written informed consent prior to the procedure using a form that is approved by the local Ethics Committee

Exclusion Criteria:

* Q-wave or non-Q-wave myocardial infarction within the preceding 72 hours unless the CK and CK-MB enzymes are back to normal
* Unprotected left main coronary disease with >= 50% stenosis
* Impaired runoff in the treatment vessel with diffuse distal disease
* Ostial target lesion
* Angiographic evidence of thrombus within target lesion
* Calcified lesions which cannot be successfully predilated
* Ejection fraction <= 30%
* Totally occluded vessel (TIMI 0 level)
* Impaired renal function (creatinine > 3.0 mg/dl)
* Pretreatment with devices other than balloon angioplasty
* Target lesion has excessive tortuosity unsuitable for stent delivery and deployment
* Target lesion involves bifurcation including a side branch >= 2.5 mm in diameter (either stenosis of both main vessel and major branch or stenosis of just major branch) that would require side branch stenting which is likely to occur if side branch is diseased and intended to be stented
* Prior stent within 5 mm of target lesion this includes in-stent restenosis
* Significant (> 50%) untreated stenoses proximal or distal to the target lesion that will not be treated during the procedure and may require revascularization or impede runoff
* Intervention of another lesion has occurred within one month before or is planned or highly probable to be performed within the next 30 days after this index procedure
* Recipient of heart transplant
* Patient with a life expectancy less than 12 months
* Known allergies to aspirin, clopidogrel bisulfate (Plavix®), ticlopidine (Ticlid®), heparin stainless steel, contrast agent, Paclitaxel or Sirolimus
* Any significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study
* Target lesion located in an arterial or venous by-pass graft
* Currently participating in an investigational drug or another device study
* Unstable angina pectoris Braunwald Classification A I-II-III or is having a peri-infarction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2004-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is angiographic in-stent late loss at 8-months follow-up as determined by quantitative coronary angiography | 8 months

SECONDARY OUTCOMES:
Target lesion and vessel revascularization (TLR, TVR) | 12 months
Major adverse cardiac events (MACE) at 30 days, 8 and 12 months | 30 days, 8 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Zehender, MD PhD, Principal Investigator — University Clinic Freiburg
Locations (1):
- Albert-Ludwig University Clinic, Freiburg im Breisgau, Baden-Wurttemberg, Germany